CLINICAL TRIAL: NCT06440265
Title: Validity and Reliability of Korean Version of Activity Measure for Post Acute Care (AM-PAC) Inpatient Short Form (Low Function) in Critically Ill Patients
Brief Title: Validity and Reliability of Korean Version of AM-PAC Inpatient Short Form (Low Function) in Critically Ill Patients
Acronym: AM-PAC
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Eun Hyun, assistant professor (MD, PhD), Department of Rehabilitation Medicine, Seoul National University Hospital
Other Study IDs: 2301-085-1395
Record Dates: First submitted 2024-04-26; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Post Intensive Care Syndrome; Intensive Care Unit Acquired Weakness
Keywords: ICU acquired weakness; Post intensive care syndrome; AM-PAC
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AM-PAC inpatient short form (low function) — The Activity Measure for Post-Acute Care(AM-PAC) "6-clicks" instruments have advantages in that they are simple and quick to complete, easy to use within usual care and has been validated in the entire hospital population. It has gained broad adoption in acute care hospital and, although it includes items for people at lower levels of function, there is a concern of a floor effect in ICU measurement. So, new AM-PAC items are developed to measure physical function at the lowest level and added 2 new items to AM-PAC inpatient mobility short form. It lowered the floor effect and increased statistical power, measurement breath, and sensitivity.
  2 new items
  * Turning head
  * Following simple instructions

SUMMARY:
The Activity Measure for Post Acute Care (AM-PAC) inpatient short form (low function) evaluates the level of assistance a patient requires another person to provide for distinct functional mobility and daily activities. The objective of the study was to translate and cross-culturally adapt the AM-PAC (low function) into Korean version and assess its reliability and validity .

Independent raters assessed 38 patients from ICU using the Korean version of AM-PAC, respectively. Intra-class correlation coefficients (ICCs) and Bland-Altman's plots were used to evaluate reliability, and Cronbach's alpha for internal consistency. Validity was evaluated using Spearman's correlation analysis with other physical function assessment tools (functional status score for the ICU(FSS-ICU), Medical Research Council-sum score(MRC-SS), hand grip strength) and other unrelated factors (body mass index, glucose level).

DETAILED DESCRIPTION:
The Activity Measure for Post Acute Care (AM-PAC) inpatient short form (low function) evaluates the level of assistance a patient requires another person to provide for distinct functional mobility and daily activities. The objective of the study was to translate and cross-culturally adapt the AM-PAC (low function) into Korean version and assess its reliability and validity.

An expert committee in intensive care unit (ICU) rehabilitation supervised the forward and backward translation process and to finalize the Korean version of AM-PAC (low function).

First evaluation of AM-PAC basic mobility and daily activity inpatient short forms was conducted on the first rehabilitation treatment day in ICU by the primary therapist. Subsequently, follow-up evaluations are conducted at 2 weeks and 4 weeks until the patient is discharged. Paired raters observed and recorded the scores independently. Each therapist was unaware of the other rater's scores, and they did not communicate verbally during the assessment. Starting with the first evaluation in the ICU, the same inter-rater reliability evaluation was performed in week 2 and week 4.

Raters assessed 38 patients from Medical ICU using the Korean version of AM-PAC. Intra-class correlation coefficients (ICCs) and Bland-Atman's plots were used to evaluate reliability, and Cronbach's alpha for internal consistency.

Then, convergent validity was evaluated using Spearman's correlation analysis between AM-PAC score and other physical function assessment tools (FSS-ICU, MRC-sum score, hand grip strength), and divergent validity was evaluated using correlation analysis between AM-PAC score and BMI or serum glucose level.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years who were admitted to the Medical ICU and were expected to remain in the ICU for at least two days, were eligible for inclusion.

Exclusion Criteria:

* Patients who were medically unstable to start rehabilitation in ICU or when mobilization was contraindicated by the medical team were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients above 18 years who were admitted to the Medical ICU and who are candidates of ICU rehabilitation, receiving the best care to recover from critical illness
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability | enrollment day, 2week, 4week
  two-way, mixed effect intra-class correlation coefficient (ICC) and Bland Altman's plot between each independent, blinded rater's AM-PAC scores
Concurrent Validity | enrollment day, 2week, 4week
  Convergent validity using Spearman's correlation analysis between AM-PAC score and FSS-ICU, MRC-sum score, hand grip strength; Divergent validity using Spearman's correlation analysis between AM-PAC score and body mass index(BMI) and serum glucose level which are irrelevant with functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Eun Hyun, MD,PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea